CLINICAL TRIAL: NCT06814899
Title: Use of Fosfomycin in the Treatment of Bacterial Infections: "real-life" Study At the ASST of Lecco
Brief Title: Use of Fosfomycin in the Treatment of Bacterial Infections
Acronym: FOSFOREAL LIFE
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Stefania Piconi, Director of Infectious Diseases Unit, Azienda Ospedaliera di Lecco
Other Study IDs: FOSFOREAL LIFE
Record Dates: First submitted 2024-05-20; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Analyze the Medical Records of Patients Admitted At ASST Lecco from 01/04/2020 to 31/12/2023 Treated with Fosfomycin IV
MeSH Terms: interventions — Fosfomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Fosfomycin — In this retrospective study, the investigators want to analyze the medical records of all patients admitted to the Lecco ASST from 04/01/2020 to 12/31/2023 treated with IV fosfomycin in order to evaluate different clinical outcomes.

SUMMARY:
Fosfomycin is an antibiotic discovered since 1969. Disodium fosfomycin, for intravenous use (C3H5Na2O4P) is a bactericidal antibiotic, available in Italy since 2019 (AIFA approval). It works by blocking the enzyme UDP-N-acetylglucosamine enolpyruvil transferase, inhibiting the synthesis of peptidoglycan. It binds poorly to plasma proteins and is distributed very well in various tissues such as: eyes, bones, skin and subcutaneous tissue, muscles, lungs, prostate, bile and inflamed meninges. It also has a strong anti-biofilm activity.

Fosfomycin is active against Gram-positive bacteria (staphylococci, streptococci, enterococci, including MRSA and VRE) and Gram-negative bacteria (Enterobacterales, Haemophilus influenzae, Proteus mirabilis, Pseudomonas aeruginosa, including MDR strains) and against difficult-to-treat bacteria such as Serratia marcescens, Stenotrophomonas maltophilia, Bacteroides spp and intracellular bacteria such as Chlamydia and Mycoplasma. It has no activity against Acinetobacter spp, Peptococcus spp. and Peptostreptococcus spp, Burkholderia cepacia, and Mycobacterium tuberculosis.

IV fosfomycin is approved for the treatment of osteomyelitis, complicated urinary tract infections, pneumonia including hospital-acquired and ventilator-associated pneumonia, complicated skin and soft tissue infections, bacterial meningitis, and complicated bacteremia.

In this retrospective study, the investigators want to analyze the medical records of all patients admitted to the ASST of Lecco from 01/04/2020 to 31/12/2023 treated with fosfomycin IV in order to evaluate different clinical outcomes given the recent introduction at ASST Lecco

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients hospitalized at A. Manzoni Lecco between April 2020 and December 2023;
* Patients treated with IV fosfomycin as monotherapy or in combination with other antibiotics for at least 72 hours.

Exclusion Criteria:

* Patients who received fosfomycin IV for less than 72h for any cause (death, adverse events, clinical decision).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at A. Manzoni Lecco between April 2020 and December 2023 and treated with IV fosfomycin as monotherapy or in combination with another antibiorics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical outcome of all patients treated with IV fosfomycin | 3 months
  Evaluation of the clinical outcome of all patients treated with IV fosfomycin intended as negative culture tests and resolution of clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefania Piconi, Lecco, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No